CLINICAL TRIAL: NCT00712855
Title: A Phase 1B, Multi-center, Open Label, Dose Escalation Study of Mapatumumab ([HGS1012], a Fully-human Monoclonal Antibody to TRAIL-R1) in Combination With Sorafenib as a First Line Therapy in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: A Study of Mapatumumab in Combination With Sorafenib in Subjects With Advanced Hepatocellular Carcinoma
Acronym: HCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGS1012-C1077
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — mapatumumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): mapatumumab and sorafenib
  Interventions: Biological: mapatumumab; Drug: sorafenib

INTERVENTIONS:
Biological: mapatumumab — 3, 10, or 30 mg/kg IV (in the vein), on day 1 of each 21 day cycle
Drug: sorafenib — 400 mg orally, twice a day continuously in each cycle
  Other Names: Nexavar

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of escalating doses of mapatumumab in combination with sorafenib in subjects with advanced Hepatocellular Carcinoma who are positive for hepatitis B surface antigen or hepatitis C antibody.

ELIGIBILITY:
Inclusion Criteria:

* Moderate liver disease
* Test positive for hepatitis B surface antigen or hepatitis C antibody
* Locally advanced unresectable/untransplantable or metastatic hepatocellular carcinoma
* Age 18 years or older

Exclusion Criteria:

* Received investigational (not yet approved by a regulatory authority) or non-investigational agent to treat hepatocellular carcinoma.
* Received radiation therapy within 4 weeks before randomization
* Major surgery within 4 weeks before randomization
* Minor surgery within 2 weeks before randomization
* Systemic steroids within 1 week before randomization
* Hepatic encephalopathy, per the investigator's evaluation
* History of clinically significant gastrointestinal bleeding requiring procedural intervention within 4 weeks before enrollment
* History of any infection requiring hospitalization or antibiotics within 2 weeks before randomization
* Known brain or spinal cord metastases
* History of other cancers within 5 years before enrollment
* Pregnant or breast-feeding women
* Known HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-06; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Type, frequency, and severity of adverse events. | Until disease progression or unacceptable toxicity develops

CONTACTS AND LOCATIONS:
Overall Officials: Norma Lynn Fox, PhD, Study Director — Human Genome Sciences Inc.
Locations (6):
- United States (6):
  - Cedars-Sinai Health System, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Pennsylvania- Abramson Cancer Center, Philadelphia, Pennsylvania